CLINICAL TRIAL: NCT02117791
Title: Drug Use Investigation of Riociguat for ChronicThromboembolic Pulmonary Hypertension (CTEPH)
Brief Title: Prospective, Non-interventional, Multi-center Post-authorization Safety Study of Riociguat for Chronic Thromboembolic Pulmonary Hypertension (CTEPH )
Acronym: JPMS-CTEPH
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16843; ADEMPAS-CTEPH (Other: company internal)
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Hypertension, Pulmonary
Keywords: Riociguat, Adempas, sGC stimulator, CTEPH, Japan, PMS
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — riociguat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Riociguat treatment group
  Interventions: Drug: Riociguat (ADEMPAS, BAY63-2521)

INTERVENTIONS:
Drug: Riociguat (ADEMPAS, BAY63-2521) — The treatment of Riociguat should comply with the local product information (start dose: 3 mg/day, maximum dose: 7.5 mg/day)

SUMMARY:
This local, prospective, non-interventional, multi-center study includes patients treated with Riociguat for inoperable CTEPH(Chronic thromboembolic pulmonary hypertension)/ persistent or recurrent CTEPH after surgical treatment. It is planned to include a total of 400 patients (valid for safety analysis). This study is performed as an all-case investigation. The treatment of Riociguat is performed based on the product label in Japan. The standard observation period is 12 months from the 1st treatment of Riociguat. Safety and effectiveness are evaluated at 4th and 12th month. In addition, the extension observation is carried out once a year for 7 years at the longest to collect information on safety and effectiveness as long as Riociguat treatment continues. When the treatment of Riociguat is terminated, observation of a patient ends. For each patient, the investigator records data as defined in the protocol at each evaluation point by using the Electronic Data Capture (EDC) system. The duration of the study is approximately 9 years from launch.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are treated with Riociguat for CTEPH

Exclusion Criteria:

* Patients who are contraindicated based on the product label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population includes patients treated with Riociguat for inoperable CTEPH/ persistent or recurrent CTEPH after surgical treatment. This study is performed as an all-case investigation. Therefore, all patients who have been treated with Riociguat for CTEPH need to be registered in principle, until the target number of patients reached.
Sampling Method: Non-Probability Sample
Enrollment: 1298 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events and adverse drug reactions | up to 8 years

SECONDARY OUTCOMES:
Change from baseline in 6MWD (6-Minute Walking Distance) after 4 and 12 months | baseline and 4 months, and 12 months
Change from baseline in Pulmonary Vascular Resistance (PVR) after 4 and 12 months | baseline and 4 months, and 12 months
Change from baseline in TRPG (Tricuspid Regurgitation Pressure Gradient) after 4 and 12 months | baseline and 4 months, and 12 months
Change from baseline in BNP/NT-pro BNP after 4 and 12 months | baseline and 4 months, and 12 months
Change from baseline in WHO (World Health Organization) functional class after 4 and 12 months | baseline and 4 months, and 12 months
Time to Clinical Worsening | up to 8 years
  The first occurrence of the following events is recorded and will be considered for the calculation of the combined endpoint: • Death (all-cause mortality) • Heart/lung transplantation • Rescue Pulmonary Endarterectomy, Rescue Balloon Pulmonary Angioplasty or Hospitalization due to persistent worsening of Pulmonary Hypertension • Start of new PH specific treatment due to worsening Pulmonary Hypertension. • Persistent decrease in 6MWD due to worsening pulmonary hypertension • Persistent worsening of functional class due to deterioration of Pulmonary Hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Tanabe N, Ogo T, Hatano M, Kigawa A, Sunaya T, Sato S. Safety and effectiveness of riociguat for chronic thromboembolic pulmonary hypertension in real-world clinical practice: interim data from post-marketing surveillance in Japan. Pulm Circ. 2020 Jul 23;10(3):2045894020938986. doi: 10.1177/2045894020938986. eCollection 2020 Jul-Sep. PMID 32754307